CLINICAL TRIAL: NCT04879745
Title: A Pilot Study of the MyVoice:Rheum Decision Aid to Address the Reproductive Health Needs of Women With Rheumatic Diseases
Brief Title: MyVoice:Rheum Decision Aid for Women With Rheumatic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Mehret Birru Talabi, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20060240; K23AR075057-01A1 (NIH)
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Results first posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Rheumatic Diseases; Physician-Patient Relations; Contraception
Keywords: rheumatic diseases; shared decision-making; sexual and reproductive health; decision aids
MeSH Terms: conditions — Rheumatic Diseases; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Aid Users (Experimental): Patients with a rheumatic disease who are given access to the MyVoice:Rheum decision aid
  Interventions: Other: MyVoice:Rheum
- Pamphlet Users (Active Comparator): Patients with a rheumatic disease who are given access to a widely-accessible pamphlet about family planning
  Interventions: Other: Pamphlet

INTERVENTIONS:
Other: MyVoice:Rheum — Participants will be given access to MyVoice:Rheum, a web-based decision aid (DA).
  Arms: Decision Aid Users
Other: Pamphlet — Participants in this arm will be given a copy of an existing patient pamphlet
  Arms: Pamphlet Users

SUMMARY:
This is a pilot trial to assess feasibility and acceptability of MyVoice:Rheum vs. a patient pamphlet among female patients ages 18-44 (n=40) who receive rheumatology care.

• Hypothesis: MyVoice:Rheum will be feasible and acceptable to patients who receive rheumatology care.

DETAILED DESCRIPTION:
The pilot will demonstrate if the MyVoice:Rheum decision aid can be feasibly and acceptably implemented into the rheumatology context and inform operational procedures for a future hybrid effectiveness-implementation trial. Women in the intervention arm will receive the MyVoice:Rheum decision aid (n=30). Women in the control arm (n=9) will receive a widely-accessible paper-based pamphlet about pregnancy, which, similarly to MyVoice:Rheum, targets women with a broad range of rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

Patients must have at least one of four rheumatic diseases diagnosed by a rheumatologist: rheumatoid arthritis (RA), systemic sclerosis (SSc), myositis, Sjogren's syndrome, vasculitis, spondyloarthritis, and systemic lupus erythematosus (SLE).

Patients must read and speak in English as a Spanish-language version of the tool has not yet been developed

Access to a smart phone, personal computer, or tablet.

Exclusion Criteria:

* Women who have had prior hysterectomy or sterilization, or are pregnant.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehret S Birru Talabi, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Falk Rheumatology Clinic, Pittsburgh, Pennsylvania
  - UPMC Lupus Center of Excellence, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta B, Luo Y, Xu J, Sammaritano L, Salmon J, Lockshin M, Goodman S, Ibrahim S. Trends in Maternal and Fetal Outcomes Among Pregnant Women With Systemic Lupus Erythematosus in the United States: A Cross-sectional Analysis. Ann Intern Med. 2019 Aug 6;171(3):164-171. doi: 10.7326/M19-0120. Epub 2019 Jul 9. PMID 31284305
- [Background] Birru Talabi M, Clowse MEB, Schwarz EB, Callegari LS, Moreland L, Borrero S. Family Planning Counseling for Women With Rheumatic Diseases. Arthritis Care Res (Hoboken). 2018 Feb;70(2):169-174. doi: 10.1002/acr.23267. No abstract available. PMID 28437837
- [Background] Rajendran A, Eudy AM, Balevic SJ, Clowse MEB. The importance of pregnancy planning in lupus pregnancies. Lupus. 2021 Apr;30(5):741-751. doi: 10.1177/0961203321989803. Epub 2021 Jan 28. PMID 33509066
- [Background] Birru Talabi M, Callegari LS, Borrero S. Redefining Primum Non Nocere to Include Reproductive Autonomy: A New Paradigm in Subspecialty Medicine. Womens Health Rep (New Rochelle). 2021 Oct 26;2(1):497-499. doi: 10.1089/whr.2021.0079. eCollection 2021. PMID 34970654
- [Background] Birru Talabi M, Eudy AM, Jayasundara M, Haroun T, Nowell WB, Curtis JR, Crow-Hercher R, White CW, Ginsberg S, Clowse MEB. Pregnancy, Periods, and "The Pill": Exploring the Reproductive Experiences of Women with Inflammatory Arthritis. ACR Open Rheumatol. 2019 Apr 15;1(2):125-132. doi: 10.1002/acr2.1016. eCollection 2019 Apr. PMID 31777789
- [Background] Stransky OM, Wolgemuth T, Kazmerski T, Chodoff A, Borrero S, Birru Talabi M. Contraception decision-making and care among reproductive-aged women with autoimmune diseases. Contraception. 2021 Feb;103(2):86-91. doi: 10.1016/j.contraception.2020.11.001. Epub 2020 Nov 9. PMID 33181126
- [Background] Wolgemuth T, Stransky OM, Chodoff A, Kazmerski TM, Clowse MEB, Birru Talabi M. Exploring the Preferences of Women Regarding Sexual and Reproductive Health Care in the Context of Rheumatology: A Qualitative Study. Arthritis Care Res (Hoboken). 2021 Aug;73(8):1194-1200. doi: 10.1002/acr.24249. Epub 2021 Jul 14. PMID 32374928
- [Background] Birru Talabi M, Clowse MEB, Blalock SJ, Hamm M, Borrero S. Perspectives of Adult Rheumatologists Regarding Family Planning Counseling and Care: A Qualitative Study. Arthritis Care Res (Hoboken). 2020 Mar;72(3):452-458. doi: 10.1002/acr.23872. PMID 30875455
- [Background] Frosch DL, Legare F, Fishbein M, Elwyn G. Adjuncts or adversaries to shared decision-making? Applying the Integrative Model of behavior to the role and design of decision support interventions in healthcare interactions. Implement Sci. 2009 Nov 12;4:73. doi: 10.1186/1748-5908-4-73. PMID 19909547
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] O'Connor AM, Llewellyn-Thomas HA, Flood AB. Modifying unwarranted variations in health care: shared decision making using patient decision aids. Health Aff (Millwood). 2004;Suppl Variation:VAR63-72. doi: 10.1377/hlthaff.var.63. PMID 15471770
- [Background] Birru Talabi M, Eudy AM, Jayasundara M, Haroun T, Nowell WB, Curtis JR, Crow-Hercher R, White W, Ginsberg S, Clowse MEB. Tough Choices: Exploring Medication Decision-Making During Pregnancy and Lactation Among Women With Inflammatory Arthritis. ACR Open Rheumatol. 2021 Jul;3(7):475-483. doi: 10.1002/acr2.11240. Epub 2021 Jun 11. PMID 34114738
- [Background] Sammaritano LR, Bermas BL, Chakravarty EE, Chambers C, Clowse MEB, Lockshin MD, Marder W, Guyatt G, Branch DW, Buyon J, Christopher-Stine L, Crow-Hercher R, Cush J, Druzin M, Kavanaugh A, Laskin CA, Plante L, Salmon J, Simard J, Somers EC, Steen V, Tedeschi SK, Vinet E, White CW, Yazdany J, Barbhaiya M, Bettendorf B, Eudy A, Jayatilleke A, Shah AA, Sullivan N, Tarter LL, Birru Talabi M, Turgunbaev M, Turner A, D'Anci KE. 2020 American College of Rheumatology Guideline for the Management of Reproductive Health in Rheumatic and Musculoskeletal Diseases. Arthritis Rheumatol. 2020 Apr;72(4):529-556. doi: 10.1002/art.41191. Epub 2020 Feb 23. PMID 32090480
- [Background] Krishnamurti T, Birru Talabi M, Callegari LS, Kazmerski TM, Borrero S. A Framework for Femtech: Guiding Principles for Developing Digital Reproductive Health Tools in the United States. J Med Internet Res. 2022 Apr 28;24(4):e36338. doi: 10.2196/36338. PMID 35482371
- [Background] Birru MS, Monaco VM, Charles L, Drew H, Njie V, Bierria T, Detlefsen E, Steinman RA. Internet usage by low-literacy adults seeking health information: an observational analysis. J Med Internet Res. 2004 Sep 3;6(3):e25. doi: 10.2196/jmir.6.3.e25. PMID 15471751
- [Background] Ng JY, Ntoumanis N, Thogersen-Ntoumani C, Deci EL, Ryan RM, Duda JL, Williams GC. Self-Determination Theory Applied to Health Contexts: A Meta-Analysis. Perspect Psychol Sci. 2012 Jul;7(4):325-40. doi: 10.1177/1745691612447309. PMID 26168470
- [Background] Torgerson DJ, Roberts C. Understanding controlled trials. Randomisation methods: concealment. BMJ. 1999 Aug 7;319(7206):375-6. doi: 10.1136/bmj.319.7206.375. No abstract available. PMID 10435967
- [Background] Birru Talabi M, Callegari LS, Kazmerski TM, Krishnamurti T, Mosley EA, Borrero S. A blueprint for a new model of sexual and reproductive health care in subspecialty medicine. Health Serv Res. 2023 Feb;58(1):216-222. doi: 10.1111/1475-6773.14074. Epub 2022 Oct 11. No abstract available. PMID 36151999
- [Background] Schwarz EB, Parisi SM, Handler SM, Koren G, Cohen ED, Shevchik GJ, Fischer GS. Clinical decision support to promote safe prescribing to women of reproductive age: a cluster-randomized trial. J Gen Intern Med. 2012 Jul;27(7):831-8. doi: 10.1007/s11606-012-1991-y. PMID 22297687
- [Background] Pryor KP, Albert B, Desai S, Ritter SY, Tarter L, Coblyn J, Bermas BL, Santacroce LM, Dutton C, Braaten KP, Pace LE, Rexrode K, Janiak E, Feldman CH. Pregnancy Intention Screening in Patients With Systemic Rheumatic Diseases: Pilot Testing a Standardized Assessment Tool. ACR Open Rheumatol. 2022 Aug;4(8):682-688. doi: 10.1002/acr2.11449. Epub 2022 May 31. PMID 35639495
- [Background] Stransky O, Hunt N, Richards JS, Talabi MB. Exploring Family Planning, Parenting, and Sexual and Reproductive Health Care Experiences of Men With Rheumatic Diseases. J Rheumatol. 2022 Mar;49(3):251-255. doi: 10.3899/jrheum.210785. Epub 2021 Nov 15. PMID 34782452
- [Background] Crear-Perry J, Hassan A, Daniel S. Advancing Birth Equity in a Post-Dobbs US. JAMA. 2022 Nov 1;328(17):1689-1690. doi: 10.1001/jama.2022.19468. PMID 36318120
- [Background] Borrero S, Talabi MB, Dehlendorf C. Confronting the Medical Community's Complicity in Marginalizing Abortion Care. JAMA. 2022 Nov 1;328(17):1701-1702. doi: 10.1001/jama.2022.18328. PMID 36318124
- [Background] Bermas BL, Blanco I, Blazer AD, Clowse ME, Edens C, Ramsey-Goldman R, Talabi MB. Overturning Roe v. Wade: Toppling the Practice of Rheumatology. Arthritis Rheumatol. 2022 Dec;74(12):1865-1867. doi: 10.1002/art.42336. Epub 2022 Oct 11. No abstract available. PMID 36128693
- [Result] Birru Talabi M, Clowse MEB, Blalock SJ, Switzer G, Yu L, Chodoff A, Borrero S. Development of ReproKnow, a reproductive knowledge assessment for women with rheumatic diseases. BMC Rheumatol. 2019 Oct 21;3:40. doi: 10.1186/s41927-019-0091-6. eCollection 2019. PMID 31660532
- [Result] Rocca CH, Ralph LJ, Wilson M, Gould H, Foster DG. Psychometric Evaluation of an Instrument to Measure Prospective Pregnancy Preferences: The Desire to Avoid Pregnancy Scale. Med Care. 2019 Feb;57(2):152-158. doi: 10.1097/MLR.0000000000001048. PMID 30550399
- [Result] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Result] Kazmerski TM, Stransky OM, Wright CE, Albanowski M, Pilewski JM, Talabi MB, Callegari LS, Chang JC, Abebe KZ, Miller E, Deal A, O'Leary R, Borrero S. Feasibility Testing of a Web-Based Reproductive Decision Support Tool for Cystic Fibrosis. J Cyst Fibros. 2024 May;23(3):404-411. doi: 10.1016/j.jcf.2023.10.003. Epub 2023 Oct 11. PMID 37833123
- [Result] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Result] Dehlendorf C, Henderson JT, Vittinghoff E, Steinauer J, Hessler D. Development of a patient-reported measure of the interpersonal quality of family planning care. Contraception. 2018 Jan;97(1):34-40. doi: 10.1016/j.contraception.2017.09.005. Epub 2017 Sep 18. PMID 28935217
- [Result] Maly RC, Frank JC, Marshall GN, DiMatteo MR, Reuben DB. Perceived efficacy in patient-physician interactions (PEPPI): validation of an instrument in older persons. J Am Geriatr Soc. 1998 Jul;46(7):889-94. doi: 10.1111/j.1532-5415.1998.tb02725.x. PMID 9670878

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decision Aid Users | Pamphlet Users
Started | 35 | 10
Post-intervention Assessment (After participants were enrolled in the study and randomized to each arm, they completed a post-intervention assessment after their visit with their rheumatologist.) | 31 | 9
Completed | 31 | 9
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid Users | Pamphlet Users | Total
Number analyzed (Participants) | 35 | 10 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 10 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 33.23 [20 to 42] | 28.80 [23 to 38] | 32.825 [20 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 10 | 45
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 32 | 10 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 28 | 7 | 35
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 10 | 45

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention
Description: Acceptability of Intervention Measure (AIM) consist of Four- item measure, Likert scales ranging from 1 (completely disagree) to 5 (completely agree). Score is determined by calculating the mean of scores, with a higher score indicating higher acceptability. We assigned a feasibility threshold of ≥ 3.5 of 5, for which higher scores indicate more positive responses.
Time Frame: T2 (within 24 hours of intervention and appointment)
Population: 30 of 31 decision aid users completed the AIM.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Aid Users | Pamphlet Users
Number analyzed (Participants) | 30 | 9
score on a scale | 4.45 (.59) | 3.97 (.65)

2. Primary Outcome: Intervention Appropriateness Measure
Description: The validated Intervention Appropriateness Measure (IAM) consist of Four-item Likert scales ranging from 1 (completely disagree) to 5 (completely agree); we assigned a feasibility threshold of ≥ 3.5 of 5 for IAM scores, for which higher scores indicate more positive responses. Score is determined by calculating the mean, with a higher score indicating greater appropriateness.
Time Frame: T2 (within 24 hours of intervention and appointment)
Population: 30 of the 31 Decision Aid users completed the IAM.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Aid Users | Pamphlet Users
Number analyzed (Participants) | 30 | 9
score on a scale | 4.48 (.61) | 4.11 (.85)

3. Primary Outcome: System Usability Scale
Description: Usability was assessed via summary scores from the System Usability Scale (SUS), which consists of a 10-item Likert scale with scores ranging from 0-100; overall score calculated by finding the mean of items on scale. We set a threshold of scores >80.3 as 'A'/excellent and 68-80.3 as 'B'/very good, consistent with standard rating for the SUS.
Time Frame: T2 (within 24 hours of intervention and appointment)
Population: 30 of the original 31 Decision Aid Users completed the SUS Measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Aid Users | Pamphlet Users
Number analyzed (Participants) | 30 | 9
score on a scale | 83.06 (15.67) | 79.32 (14.10)

4. Other Pre Specified Outcome: Reproductive Knowledge Assessment for Women With Rheumatic Diseases (ReproKnow)
Description: Rheumatology-specific reproductive health knowledge was assessed via ReproKnow, a measure developed and preliminarily validated by our team that covers domains of contraception safety and efficacy, pregnancy management, pre-conception planning, medication safety, fertility; a score of nine indicates the highest level of reproductive knowledge
Time Frame: T2 (within 24 hours of intervention and appointment) compared to T0 (baseline)
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | Decision Aid Users | Pamphlet Users
Number analyzed (Participants) | 31 | 9
number of correct responses
  T2 | 7.27 (1.17) | 7.11 (2.50)
  T0 | 5.77 (1.76) | 5.44 (2.74)

5. Other Pre Specified Outcome: Perceived Efficacy in Patient-Physician Interactions
Description: Self-reported efficacy in communicating with providers was assessed using a modified version of the validated five-item Perceived Efficacy in Patient-Provider Interactions (PEPPI) scale. Five-item measure with 5-point Likert scale questions from 1 (not at all confident) to 5 (very confident). Aggregate score is calculated by taking the individual item scores together and dividing by 5, with higher score indicating higher perceived efficacy in communicating with providers.
Time Frame: T2 (within 24 hours of intervention and appointment) compared to T0 (baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Aid Users | Pamphlet Users
Number analyzed (Participants) | 31 | 9
score on a scale
  T2 | 4.07 (0.82) | 3.98 (.98)
  T0 | 3.47 (1.19) | 3.73 (.92)

6. Other Pre Specified Outcome: Participant Number of Pregnancies During Study
Description: Assessed by participant-reported survey responses to a Yes/No item about whether a pregnancy has occurred since enrollment.
Time Frame: T3 (three months post-intervention)
Population: Pamphlet users did not complete T3 assessment. 30 Decision aids users completed T3 assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid Users | Pamphlet Users
Number analyzed (Participants) | 30 | 0
Participants
  Pregnant | 1 | 0
  Not pregnant | 29 | 0

7. Other Pre Specified Outcome: Quantity and Quality of Reproductive Health Conversation With Rheumatologist
Description: Three-item measure. Did you talk to your rheumatologist about family planning today- yes/no; Did you make a decision related to family planning- yes/no; what was the family planning decision you made today? (Not Reported)
Time Frame: T2 (within 24 hours of intervention and appointment)
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid Users | Pamphlet Users
Number analyzed (Participants) | 31 | 9
Participants
  Did you talk to your Rheumatologist today about family planning?: Yes | 17 | 4
  Did you talk to your Rheumatologist today about family planning?: No | 14 | 5
  Did you make a decision related to family planning?: Yes | 6 | 1
  Did you make a decision related to family planning?: No | 25 | 8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Decision Aid Users | Pamphlet Users
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/10
Other Adverse Events (participants affected / at risk) | 0/31 | 0/10

LIMITATIONS AND CAVEATS:
Due to an increase in telemedicine utilization over the COVID-19 pandemic, most recruitment was conducted remotely instead of in-person as originally intended. The COVID-19 pandemic coincided with our study, which may account for the low number of participants recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT04879745/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT04879745/ICF_001.pdf